CLINICAL TRIAL: NCT04486482
Title: An Exploratory, Open Label, Clinical Study to Evaluate the Physiologic Effects of KB109 in Adult Patients With Mild-to-Moderate COVID-19 on Gut Microbiota Structure and Function in the Outpatient Setting
Brief Title: A Clinical Study to Assess the Physiologic Effects of KB109 in Patients With COVID-19 on Gut Microbiota Structure and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaleido Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K032-120
Record Dates: First submitted 2020-07-23; First posted 2020-07-24 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Mild-to-Moderate COVID-19
Keywords: Microbiome; COVID-19; Corona Virus; Corona Virus Disease; Kaleido; Kaleido Biosciences; KB109; Oligosaccharides; Glycan; Outpatient; Pathogens; Microbiome Metabolic Therapy; MMT; Telemedicine
MeSH Terms: conditions — COVID-19 | interventions — Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KB109 + Self Supportive Care (SSC) (Other)
  Interventions: Other: KB109 + Self Supportive Care (SSC)
- Self Supportive Care (SSC) Alone (Other)
  Interventions: Other: Self Supportive Care (SSC) Alone

INTERVENTIONS:
Other: KB109 + Self Supportive Care (SSC) — KB109 is a novel glycan
  Arms: KB109 + Self Supportive Care (SSC)
Other: Self Supportive Care (SSC) Alone — Self Supportive Care (SSC) Alone
  Arms: Self Supportive Care (SSC) Alone

SUMMARY:
This exploratory, open-label clinical study aims to explore the physiologic effects of KB109, a novel glycan, on adult patients with COVID-19 illness on gut microbiota structure and function in the outpatient setting.

ELIGIBILITY:
To be considered for enrollment into this study, each patient must meet all of the following Inclusion Criteria:

1. Be male or female, ≥18 years of age
2. Be willing and able to give informed consent
3. Screening/Randomization telemedicine visit within 2 days of testing positive test for COVID-19
4. Having self-reported fever or cough for not more than 72 hours prior to COVID-19 testing
5. Mild to moderate COVID-19
6. Able to adhere to the study visit schedule and other protocol requirements

Patients who meet any of the following Exclusion Criteria at the Randomization Visit will not be enrolled into the study:

1. Patients who are hospitalized for in-patient treatment or currently being evaluated for potential hospitalization at the time of informed consent for conditions other than COVID-19
2. History of chronic lung disease
3. Ongoing requirement for oxygen therapy
4. Shortness of breath in resting position
5. Diagnosis of sleep apnea requiring Bilevel Positive Airway Pressure (BIPAP) / Continuous Positive Airway Pressure (CPAP)
6. Female patients who are pregnant, trying to become pregnant or lactating.
7. Is considered, in the opinion of the PI, to be unlikely for any reason to be able to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing study-product related treatment-emergent adverse events (TEAEs) | Day 1 to Day 35

SECONDARY OUTCOMES:
Relative abundance of microbial taxa in fecal samples as assessed by shotgun profiling based on shotgun sequencing. | Day 1 to Day 35
  Change from baseline in relative abundance of microbial taxa (operational taxanomic units) in the KB109 + SSC group versus SSC alone

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wingertzahn, PhD, Study Director — Kaleido Biosciences
Locations (12):
- United States (12):
  - Cullman Clinical Trials, Cullman, Alabama
  - American Institute of Research, Los Angeles, California
  - Rancho Cucamonga Clinical Research, Rancho Cucamonga, California
  - Next Phase Research Alliance, Boca Raton, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Hope Clinical Trials, Miami, Florida
  - Kendall South Medical Center, Inc., Miami, Florida
  - Quad Clinical Research, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Inquest Research, Baytown, Texas
  - Olympus Family Medicine, Salt Lake City, Utah
  - South Ogden Family Medicine Center, South Ogden, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haran JP, Pinero JC, Zheng Y, Palma NA, Wingertzahn M. Virtualized clinical studies to assess the natural history and impact of gut microbiome modulation in non-hospitalized patients with mild to moderate COVID-19 a randomized, open-label, prospective study with a parallel group study evaluating the physiologic effects of KB109 on gut microbiota structure and function: a structured summary of a study protocol for a randomized controlled study. Trials. 2021 Apr 2;22(1):245. doi: 10.1186/s13063-021-05157-0. PMID 33810796